CLINICAL TRIAL: NCT05911477
Title: Effect of rhBMP-2 on Early Bone Formation in Patients With Osteoporosis After Lumbar Fusion
Brief Title: Recombinant Human Bone Morphogenetic Protein-2(rhBMP-2) in Patients With Osteoporosis After Lumbar Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Hu Xueyu, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20222249-1
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis; Spinal Fusion
Keywords: rhBMP-2, lumbar fusion, fusion rate, osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rhBMP-2 group (Experimental)
  Interventions: Drug: RhBMP-2
- No rhBMP-2 group (No Intervention)

INTERVENTIONS:
Drug: RhBMP-2 — 1mg RhBMP-2 for one fusion-level
  Arms: rhBMP-2 group

SUMMARY:
rhBMP-2 has been used to promote spinal fusion. Despite potential risk of complications, satisfied results could be obtained with low dose of rhBMP-2. Effect of early bone formation has been validated using rat ovariectomy osteoporosis model. However, whether it functioned in patients with osteoporosis remained unknown. In this study, the investigators intend to investigate whether rhBMP-2 promotes early bone formation in patients with osteoporosis after transforaminal lumbar interbody fusion (TLIF).

DETAILED DESCRIPTION:
Pseudoarthrosis and many complications associated with iliac crest bone graft (ICBG) has prompted the spine surgeons to seek alternative methods to promote rate of spinal fusion. The rhBMP-2 received FDA approval in 2002 for use as an alternative to autograft for single-level anterior lumbar interbody fusion (ALIF). Many studies reported equivalent or better fusion rates. Recent studies, however, identified complications related to rhBMP-2 use such as osteolysis, graft subsidence, and retrograde ejaculation and other urological complications. Overdose of rhBMP-2 in patients may lead to complications mentioned above. A recent randomized controlled trial in 2022 confirmed a low dose usage of rhBMP-2 promoted fusion after TLIF (21.mg per fusion level) without increase in complications.

Current fusion methods achieve interbody fusion by filling the cage in the central region of the intervertebral space with bone graft material. However, the early fusion rates (at 3 and 6 months postoperatively) are often unsatisfactory. According to present literatures, the 3-month and 6-month fusion rates have ranged from 2.9% to 43.1% and 30% to 68.8%, respectively. Although a lack of fusion may be asymptomatic, it may potentially lead to complications, even a reoperation. In addition, failure to achieve early fusion may result in a delayed return to work, and reduced patient satisfaction, especially in patients with osteoporosis. Whether rhBMP-2 may lead to higher and early fusion rate in osteoporosis patient remains unknown.

In this study, the investigators intend to compare the time it takes to achieve osseous union/fusion and the clinical efficacy of using rhBMP-2 to control group in TLIF. The rhBMP-2 in the study is produced by a domestic enterprise (HANGZHOU JIUYUAN GENE ENGINEERING CO .,LTD., Hangzhou, China).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with degenerative lumbar diseases.
* patients underwent one-level TLIF
* osteoporosis (DXA T≤-2.5)
* complete preoperative and follow-up data (imaging and health-related quality of life)

Exclusion Criteria:

* history of previous spinal surgery
* inflammatory and neoplastic diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Fusion rate at 6 months | 6 months follow-up
  1. <5°of angular motion, ≤3 mm of translation from lumbar spine dynamic radiographs
  2. Bridging bone connecting the adjacent vertebral bodies either through the implants or around the implants, and an absence of radiolucent lines around >50% of either implant from computed tomography (CT) scans of lumbar
Fusion rate at 3 months | 3 months follow-up
  <5°of angular motion, ≤3 mm of translation from lumbar spine dynamic radiographs of radiolucent lines around >50% of either implant

SECONDARY OUTCOMES:
Visual Analog Score for low back pain (VAS-B) | pre- and post-operative immediately, 3- and 6- months follow-up
  range from 0-10, a higher score means a worse outcome.Short Form Survey (SF-36)
Visual Analog Score for leg pain (VAS-L) | pre- and post-operative immediately, 3- and 6- months follow-up
  range from 0-10, a higher score means a worse outcome.
Oswestry disability index (ODI) | pre-operatively, 3- and 6-months follow-up
  range from 0-100%, a higher score means a worse outcome.
36-Item Short Form Survey (SF-36) | pre-operatively, 3- and 6-months follow-up
  As part of the Medical Outcomes Study (MOS), a multi-year, multi-site study to explain variations in patient outcomes, RAND developed the 36-Item Short Form Health Survey (SF-36) in 1992. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
Incidence of complications | post-operative immediately, 3- and 6- months follow-up
  infection, revision surgery, etc.

IPD SHARING:
Plan to Share IPD: Yes
Other researchers should ask for permissions from the investigator.
Supporting Information: Study Protocol, SAP
Time Frame: one year after the study is finished.
Access Criteria: Through emails after Obtaining written permission from the investigator